CLINICAL TRIAL: NCT01388140
Title: A Psychopathological Study of Dissociative Disorders in Psychiatric Inpatients at an Acute Stage
Brief Title: Psychopathology of Dissociative Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hai-Gwo Hwu, Visiting physician, Professor, National Taiwan University Hospital
Other Study IDs: 201012003RB
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-01

CONDITIONS: Dissociative Disorders
Keywords: dissociation; psychosis; trauma; parenting; executive functions
MeSH Terms: conditions — Dissociative Disorders; Psychotic Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- psychiatric inpatients, regardless of clinical diagnoses

SUMMARY:
The goal of the project is to investigate the prevalence of dissociative disorders in psychiatric inpatients in Taiwan. Relevant clinical issues, including common psychiatric comorbidity (e.g., positive psychotic symptoms), associated psychosocial factors (e.g., negative life events, perceived parenting style), and neuro-cognitive underpinning (e.g., executive functions) were also targeted. Standardized interview schedules, self-report scales, and cognitive tasks will be applied. The investigators hypothesized that dissociative disorders would be associated with positive psychotic symptoms, a history of early interpersonal adversity, and enhanced executive functions.

DETAILED DESCRIPTION:
Though formally included in the Diagnostic and Statistic Manual of Mental Disorders since 1980, dissociation had once been considered as a rare psychiatric disturbance. With standardized structured interview, however, recent empirical studies showed that in average 9 percent of participants in general population, 10 percent in psychiatric outpatients, and 15 percent in psychiatric inpatients receive the diagnosis of a dissociative disorder. In Taiwan few attempts have been made for systematic investigation of dissociative disorders. Little has been known about the characteristics, prevalence, and associated features of Taiwanese patients with a dissociative disorder. The goal of the project is to investigate the prevalence of dissociative disorders in psychiatric inpatients in Taiwan. Relevant clinical issues, including common psychiatric comorbidity (e.g., positive psychotic symptoms), associated psychosocial factors (e.g., negative life events, perceived parenting style), and neuro-cognitive underpinning (e.g., executive functions) were also targeted. Standardized interview schedules, self-report scales, and cognitive tasks will be applied and the assessment will be held by the licensed clinical psychologist who receive training on the assessment and treatment of dissociative disorders. The results may enhance the understanding about the clinical features of dissociative disorders in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* being stable and appropriate for interviews

Exclusion Criteria:

* with organic syndromes
* mentally retarded (FIQ <80)
* cannot communicate in Mandarin Chinese

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: psychiatric inpatients in a acute stage
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Xiao Z, Yan H, Wang Z, Zou Z, Xu Y, Chen J, Zhang H, Ross CA, Keyes BB. Trauma and dissociation in China. Am J Psychiatry. 2006 Aug;163(8):1388-91. doi: 10.1176/ajp.2006.163.8.1388. PMID 16877651
- [Background] Draijer N, Langeland W. Childhood trauma and perceived parental dysfunction in the etiology of dissociative symptoms in psychiatric inpatients. Am J Psychiatry. 1999 Mar;156(3):379-85. doi: 10.1176/ajp.156.3.379. PMID 10080552
- [Background] Chiu CD, Yeh YY, Huang YM, Wu YC, Chiu YC. The set switching function of nonclinical dissociators under negative emotion. J Abnorm Psychol. 2009 Feb;118(1):214-22. doi: 10.1037/a0014654. PMID 19222327